CLINICAL TRIAL: NCT06633419
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Effects of Multiple Doses of Carbamazepine on the Single-Dose Pharmacokinetics of MK-5684 in Healthy Adult Male Participants
Brief Title: A Drug-Drug Interaction Study of Carbamazepine and Opevesostat (MK-5684) in Healthy Adult Male Participants (MK-5684-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 5684-012; MK-5684-012 (Other: MSD)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — Prednisone; fludrocortisone acetate; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Opevesostat Period 1 (Experimental): On Day 1 a single dose of opevesostat will be administered under fasting conditions and a single dose of hormone replacement therapy (HRT) (prednisone and fludrocortisone) will be administered under fed conditions approximately 4.5 hours after opevesostat dosing.
  Interventions: Drug: Opevesostat; Drug: Prednisone; Drug: Fludrocortisone acetate
- Opevesostat Period 2 (Experimental): There will be a washout of at least 5 days between opevesostat dosing in Period 1 and the first carbamazepine dosing in Period 2. In Period 2, carbamazepine will be administered twice daily (BID) for 17 consecutive days with a single dose of opevesostat coadministered on the morning of Day 14 under fasting conditions. HRT (prednisone and fludrocortisone) will be administered under fed conditions on Day 14, approximately 4.5 hours after opevesostat and/or carbamazepine dosing.
  Interventions: Drug: Opevesostat; Drug: Prednisone; Drug: Fludrocortisone acetate; Drug: Carbamazepine

INTERVENTIONS:
Drug: Opevesostat — Administered via oral tablet per dosing regimen.
  Other Names: MK-5684; ODM-208
Drug: Prednisone — Administered at a dose of 5 mg or 10 mg dependent on HRT dosing regimen via oral tablets.
  Other Names: RAYOS®; STERAPRED®; DELTASONE®
Drug: Fludrocortisone acetate — Administered at a dose of 0.05 mg or 0.1 mg dependent on HRT dosing regimen via oral tablets.
  Other Names: FLORINEF®
Drug: Carbamazepine — Administered at a dose of 100 mg, 200 mg, or 300 mg BID dependent on dosing regimen via oral capsule (extended-release).
  Other Names: TEGRETOL®
  Arms: Opevesostat Period 2

SUMMARY:
Researchers have designed a study medicine called opevesostat as a new way to treat prostate cancer.

The purpose of this study is to learn what happens to opevesostat in a person's body over time (a pharmacokinetic or PK study). Researchers will compare what happens to opevesostat in the body when it is given with and without another medicine called carbamazepine.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m^2
* Able to swallow multiple tablets

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History or presence of any of the following:

  * Adrenal insufficiency
  * Hepatic or renal impairment
  * Gallstones, hepatitis disease, or hepatic porphyrias
  * Psychosis
  * Clinically significant hypotension, cardiac arrhythmia, cardiac conduction abnormalities, or recurrent unexplained syncopal events
  * Second- or third-degree atrioventricular heart block
  * Clinically significant sick sinus syndrome
  * Recurrent seizures, increased risk for seizures, or myasthenia gravis
  * Clinically significant hematologic disorders/blood dyscrasias, including adverse hematologic reactions to any drugs or experimental therapies
  * Any systemic fungal infection
  * Chronic infection
  * Glaucoma
  * Hypothyroidism
  * Unexplained electrolyte abnormalities, current hyponatremia, diuretic use, or syndrome of inappropriate antidiuretic hormone secretion (siADH)
  * Severe dermatologic reaction
  * Stomach ulcer
* Has a first-degree relative with multiple unexplained syncopal events, unexplained cardiac arrest, or sudden cardiac death, or has a known family history of an inherited arrhythmia syndrome (including Brugada syndrome)
* History of cancer (malignancy)
* Unable to refrain from or anticipates the use of: Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from 0 to infinity after single dosing (AUC0-inf) of opevesostat in plasma | Predose, and at designated timepoints up to 96 hours post-dose
  AUC0-inf of opevesostat in plasma will be determined.
Area under the concentration versus time curve from 0 to last quantifiable sample (AUC0-last) of opevesostat in plasma | Predose, and at designated timepoints up to 96 hours post-dose
  AUC0-last of opevesostat in plasma will be determined.
Area under the concentration versus time curve from 0 to hour 24 (AUC0-24) of opevesostat in plasma | Predose, and at designated timepoints up to 24 hours post-dose
  AUC0-24 of opevesostat in plasma will be determined.
Maximum concentration (Cmax) of opevesostat in plasma | Predose, and at designated timepoints up to 96 hours post-dose
  Cmax of opevesostat in plasma will be determined.
Time to Maximum concentration (Tmax) of opevesostat in plasma | Predose, and at designated timepoints up to 96 hours post-dose
  Tmax of opevesostat in plasma will be determined.
Apparent terminal half-life (t1/2) of opevesostat in plasma | Predose, and at designated timepoints up to 96 hours post-dose
  t1/2 of opevesostat in plasma will be determined.
Apparent Clearance (CL/F) of opevesostat in plasma | Predose, and at designated timepoints up to 96 hours post-dose
  CL/F of opevesostat in plasma will be determined.
Apparent volume of distribution during terminal phase (Vz/F) of opevesostat in plasma | Predose, and at designated timepoints up to 96 hours post-dose
  Vz/F of opevesostat in plasma will be determined.

SECONDARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to approximately 49 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be determined.
Number of participants who discontinue study intervention due to an AE | Up to approximately 49 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue from the study due to an AE will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/